CLINICAL TRIAL: NCT00314145
Title: A Multicentre, Randomized, Double-blind, Phase III Study of The Comparative Immunogenicity, Safety and Tolerability of Two Japanese Encephalitis Vaccines (ChimeriVax™-JE and JE-VAX®)
Brief Title: A Safety and Efficacy Study of Two Japanese Encephalitis Vaccines ChimeriVax™-JE and JE-VAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-009
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChimeriVax™-JE (Experimental): Participants received dose each of saline placebo on Days 0 and 7. On Day 30, participants received vaccinations of ChimeriVax™-JE vaccine and saline placebo into different arms.
  Interventions: Biological: ChimeriVax™-JE
- JE-VAX® (Active Comparator): Participants received 1 dose each of JE-VAX® vaccine on Days 0, 7, and 30, and a dose of saline placebo into a different arm on Day 30.
  Interventions: Biological: JE-VAX®

INTERVENTIONS:
Biological: ChimeriVax™-JE — 0.5 mL, Subcutaneous (ChimeriVax™-JE); 1.0 mL, (Saline)
  Arms: ChimeriVax™-JE
Biological: JE-VAX® — 0.5 mL, Subcutaneous (JE-Vax®); 1.0 mL, (Saline)
  Arms: JE-VAX®

SUMMARY:
The purpose of this study is to determine non-inferiority in seroconversion and to compare the safety and tolerability between ChimeriVaxTM-JE and JE-VAX to the respective homologous virus strain after completion of vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or above
* Subjects in good general health.
* Females must have negative pregnancy test and be using adequate form of contraception

Exclusion Criteria:

* History of vaccination/infection with JE or Yellow fever or other flaviviruses
* History of residence/travel to flavivirus endemic regions
* History of anaphylaxis/serious adverse reactions
* Administration of vaccine within 30 days of study or during treatment period
* Clinically significant physical exam/medical history/lab abnormalities
* Pregnancy
* Excessive alcohol/drug abuse
* Hypersensitivity to constituents of JE-VAX®
* Blood transfusion/treatment with blood product within 6months of study and during study treatment period
* Known/suspected immunodeficiency
* Compromised blood brain barrier
* Employees of Clinical Research Organization (CRO)/study site staff
* Any other condition which would exclude subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angles, M.D., Principal Investigator — Heart of America Research Institute
Locations (10):
- United States (5):
  - Chicago, Illinois
  - Shawnee Mission, Kansas
  - Missoula, Montana
  - Dallas, Texas
  - Tacoma, Washington
- Australia (5):
  - Adelaide
  - Melbourne
  - New South Wales
  - Queensland
  - Victoria

REFERENCES:
- [Derived] Torresi J, McCarthy K, Feroldi E, Meric C. Immunogenicity, safety and tolerability in adults of a new single-dose, live-attenuated vaccine against Japanese encephalitis: Randomised controlled phase 3 trials. Vaccine. 2010 Nov 23;28(50):7993-8000. doi: 10.1016/j.vaccine.2010.09.035. Epub 2010 Oct 8. PMID 20934459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 07 November 2005 to 15 November 2006 at 5 clinical centers in Australia and 5 clinical centers in the US.
Pre-assignment Details: A total of 820 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- JE-VAX®: All participants received 1 subcutaneous dose each of JE-VAX® vaccine on Days 0, 7, and 30, and a subcutaneous dose of saline placebo into a different arm on Day 30.
- ChimeriVax™-JE: All participants received 1 dose each of saline placebo on Days 0 and 7. On Day 30, participants received vaccinations of ChimeriVax™-JE vaccine 4 log10 Plaque-forming unit (PFU) and saline placebo into different arms.
Period: Overall Study
Arm/Group | JE-VAX® | ChimeriVax™-JE
Started | 410 | 410
Completed | 389 | 381
Not Completed | 21 | 29
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Lost to Follow-up | 5 | 12
Not completed — Physician Decision | 3 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — Sponsor Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JE-VAX® | ChimeriVax™-JE | Total
Number analyzed (Participants) | 410 | 410 | 820
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 410 | 410 | 820
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (14.81) | 37.7 (15.11) | 37.4 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 217 | 422
  Male | 205 | 193 | 398
Region of Enrollment [Number; unit: Participants]
  Australia | 203 | 120 | 323
  United States | 207 | 290 | 497

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Japanese Encephalitis (Homologous Virus) Seroconversion Following Either ChimeriVax™-JE or JE-Vax® Vaccination
Description: Antibodies to Japanese encephalitis (JE) were measured by 50% plaque reduction neutralization test (PRNT50). Seroconversion was defined as a titer of ≥ 1:10.
Time Frame: Up to Day 60 post-first vaccination
Population: Seroconversion was assessed in all participants who were seronegative to JE (both Nakayama and ChimeriVax™-JE strains) at baseline and had no protocol violations that would have interfered with evaluation of primary outcomes (Efficacy Population).
Measure: Number; unit: Participants
Groups:
- ChimeriVax™-JE: All participants received 1 subcutaneous dose each of saline placebo on Days 0 and 7. On Day 30, participants received vaccinations of ChimeriVax™-JE vaccine 4 log10 PFU and saline placebo into different arms.
Arm/Group | JE-VAX® | ChimeriVax™-JE
Number analyzed (Participants) | 365 | 346
Participants
  Day 44 (N = 0, 346) | NA — Seroconversion was not assessed at this time point for this group. | 324
  Day 60 (N = 365, 346) | 273 | 343

2. Secondary Outcome: Neutralizing Antibody Geometric Mean Titers (GMTs) to Japanese Encephalitis (Homologous Virus) Following Either ChimeriVax™-JE or JE-Vax® Vaccination
Description: Antibodies to Japanese encephalitis (JE) were measured by 50% plaque reduction neutralization test (PRNT50).
Time Frame: Up to Day 60 post-first vaccination
Population: Geometric mean titers were assessed in all participants who were seronegative to JE (both Nakayama and ChimeriVax™-JE strains) at baseline and had no protocol violations that would have interfered with evaluation of primary outcomes (Efficacy Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | JE-VAX® | ChimeriVax™-JE
Number analyzed (Participants) | 365 | 346
Titers
  Day 44 (N = 0, 346) | NA [NA to NA] — Geometric mean titers were not assessed at this time point for this group. | 312.3 [255.1 to 382.3]
  Day 60 (N = 365, 346) | 37.4 [32.5 to 42.9] | 1391.7 [1156.6 to 1674.5]

3. Secondary Outcome: Number of Participants in the Japanese Encephalitis (Homologous Virus) Neutralizing Antibody Titer Categories on Day 60 Following Either ChimeriVax™-JE or JE-Vax® Vaccination
Description: Antibodies to Japanese encephalitis (JE) were measured by 50% plaque reduction neutralization test (PRNT50).
Time Frame: Day 60 post-first vaccination
Population: Antibody titers were assessed in all participants who were seronegative to JE (both Nakayama and ChimeriVax™-JE strains) at baseline and had no protocol violations that would have interfered with evaluation of primary outcomes (Efficacy Population).
Measure: Number; unit: Participants
Arm/Group | JE-VAX® | ChimeriVax™-JE
Number analyzed (Participants) | 365 | 346
Participants
  Titer < 10 | 63 | 3
  Titer 10 to < 20 | 29 | 0
  Titer 20 to < 40 | 51 | 4
  Titer 40 to < 160 | 151 | 18
  Titer 160 to < 640 | 63 | 76
  Titer 640 to < 2560 | 6 | 75
  Titer ≥ 2560 | 2 | 170

4. Primary Outcome: Number of Participants Reporting Treatment Emergent Local Adverse Events and Treatment Emergent Systemic Reactions Post-Vaccination With Either ChimeriVax™-JE or JE-Vax®
Description: Treatment emergent local adverse events: Pain, Erythema, Pruritus, Swelling, Induration, and others as reported.
  Treatment emergent systemic reactions: Fatigue, Malaise, Chills, Pyrexia, Headache, Myalgia, Arthralgia, Diarrhea, Nausea, Vomiting, and Rash.
Time Frame: Day 0 (Pre-vaccination) up to 60 days post-first vaccination
Population: Treatment emergent local adverse events and systemic reactions were assessed in all subjects who had at least one injection (ChimeriVax™-JE, JE-Vax®, or placebo), according to the treatment actually received (Safety Population).
Measure: Number; unit: Participants
Arm/Group | JE-VAX® | ChimeriVax™-JE
Number analyzed (Participants) | 410 | 410
Participants
  Injection Site Pain | 262 | 105
  Injection Site Erythema | 123 | 27
  Injection Site Pruritus | 107 | 29
  Injection Site Swelling | 85 | 15
  Injection Site Hemorrhage | 20 | 14
  Injection Site Rash | 6 | 2
  Injection Site Edema | 2 | 0
  Injection Site Joint Pain | 1 | 1
  Injection Site Reaction | 1 | 1
  Injection Site Discomfort | 1 | 0
  Injection Site Joint Movement Impairment | 0 | 1
  Injection Site Warmth | 0 | 1
  Venipuncture Site Bruise | 1 | 0
  Fatigue | 131 | 152
  Malaise | 113 | 113
  Chills | 32 | 43
  Pyrexia | 18 | 14
  Headache | 190 | 193
  Myalgia | 107 | 105
  Arthralgia | 58 | 58
  Diarrhea | 56 | 57
  Nausea | 53 | 56
  Vomiting | 15 | 13
  Rash | 26 | 23

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) through Day 60 post first vaccination.
Arm/Group | JE-VAX® | ChimeriVax™-JE
Serious Adverse Events (participants affected / at risk) | 3/410 | 2/410
Other Adverse Events (participants affected / at risk) | 262/410 | 193/410
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-VAX® (N=410) | ChimeriVax™-JE (N=410)
Non Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE-VAX® (N=410) | ChimeriVax™-JE (N=410)
Diarrhea (Gastrointestinal disorders) | 56 (80) | 57 (99)
Nausea (Gastrointestinal disorders) | 53 (96) | 56 (75)
Chills (General disorders) | 32 (48) | 43 (68)
Fatigue (General disorders) | 131 (399) | 152 (366)
Injection Site Pain (General disorders) | 262 (804) | 105 (207)
Injection Site Erythema (General disorders) | 123 (256) | 27 (35)
Injection Site Pruritus (General disorders) | 107 (187) | 29 (46)
Injection Site Swelling (General disorders) | 85 (149) | 15 (16)
Malaise (General disorders) | 113 (248) | 113 (224)
Myalgia (Musculoskeletal and connective tissue disorders) | 107 (228) | 105 (192)
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 (99) | 58 (122)
Headache (Nervous system disorders) | 190 (546) | 193 (465)
Rash (Skin and subcutaneous tissue disorders) | 26 (36) | 23 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.